CLINICAL TRIAL: NCT04385342
Title: Follicle Stimulating Hormone (FSH) Followed by Human Menopausal Gonadotropin (HMG) Versus FSH Plus HMG During Controlled Ovarian Stimulation for in Vitro Fertilization
Brief Title: FSH Followed by HMG vs FSH Plus HMG in IVF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R.20.04.823
Record Dates: First submitted 2020-01-10; First posted 2020-05-12 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: IVF
Keywords: ovarian stimulation; subfertility; FSH; HMG
MeSH Terms: conditions — Infertility | interventions — follitropin alfa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FSH then HP-hMG (Active Comparator): Women will receive 225 IU FSH alone from day one of ovarian stimulation and when the follicular diameters reaches 10-12 mm, the 150 IU HP-hMG will substitute FSH and continued to the day of triggering
  Interventions: Drug: FSH; Drug: HP-hMG
- FSH + HP-hMG (Active Comparator): Women will receive 150 IU FSH plus 75IU HP-hMG from day one of ovarian stimulation and when the follicular diameters reaches 10-12 mm 150 IU HP-HMG till day of triggering
  Interventions: Drug: FSH; Drug: HP-hMG

INTERVENTIONS:
Drug: FSH — Controlled ovarian stimulation by FSH followed by HMG versus FSH plus HMG
  Other Names: Fostimon, Gonal-F, Puragon
Drug: HP-hMG — Controlled ovarian stimulation by FSH followed by HMG versus FSH plus HMG
  Other Names: Meriofert, Menopure

SUMMARY:
The aim of this study is to compare the clinical outcomes of sequential administration of FSH and HP-hMG FSH alone versus concomitant administration of FSH and HP-hMG during controlled ovarian stimulation in IVF cycles.

DETAILED DESCRIPTION:
Women who are planned to be subjected to IVF/ICSI through COS by long GnRHa protocol will be assessed for possibility of participation in our study. Eligible participants in our study will be those with regular menstrual cycle (21-35 days) and normal uterine anatomy (confirmed by transvaginal ultrasound examination and in some cases hysteronsalpingography and hysteroscopy).

Women with any of the following criteria will be excluded from the study: 1) age < 20 or > 37 years; 2) body mass index (BMI) < 18 or > 25 kg/m2; 3) low ovarian reserve (AFC < 7 and/or AMH < 1.1 ng/ml); 4) presence of polycystic ovarian syndrome (PCOS), endometrioma or hydrosalpinx; 5) history of chemotherapy, radiotherapy or ovarian surgery; 6) the husband needs testicular biopsy to obtain sperm; or 7) previous implantation failure.

A written informed consent will be taken from each women selected to participate before inclusion in the study. All women participating in the study will start GnRHa on day 21 of the preceding cycle and when down regulation occurs each woman will be randomly allocated into one of the two groups; group 1 and group 2. Women in group 1 will receive 225 IU FSH alone from day one of ovarian stimulation and when the follicular diameters reaches 10-12 mm, the 150 IU HP-hMG will substitute FSH and continued to the day of triggering. Women in group 2 will receive 150 IU FSH plus 75 IU HP-hMG from day one of ovarian stimulation and 150IU HP-HMG when the follicular diameters reaches 10-12 mm till day of triggering. The randomization will be simple and balanced (1:1) and will be carried out by a nurse through sealed, unlabeled, opaque envelopes containing computer-generated random numbers. The data assesor will be blinded to group assignment.

In both groups, estradiol and LH will be measured on the third day of menstruation before start of stimulation and on day 6 of stimulation TVS will be performed. Progesterone and E2 will be measured and on day of triggering. The primary outcome measure of this study will be the ongoing pregnancy rate. The secondary outcomes measures will be cancellation rate, the number of oocytes retrieved, the number of embryos, the number of vitrified embryos, the clinical pregnancy rate, the implantation rate, OHSS rate, multiple pregnancy rate, and the miscarriage rate.

ELIGIBILITY:
Inclusion Criteria:

* Women who are planned to be subjected to IVF/ICSI through COS by long GnRHa protocol.
* Women with regular menstrual cycle (21-35 days) and normal uterine anatomy (confirmed by transvaginal ultrasound examination and in some cases hysteronsalpingography and hysteroscopy).

Exclusion Criteria:

* Age < 20 or > 37 years.
* Body mass index (BMI) < 18 or > 30 kg/m2.
* Low ovarian reserve (AFC < 7 and/or AMH < 1.1 ng/ml).
* Presence of polycystic ovarian syndrome (PCOS).
* Endometrioma or hydrosalpinx.
* History of chemotherapy, radiotherapy or ovarian surgery.
* The husband needs testicular biopsy to obtain sperm.
* Previous implantation failure.

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 530 (Estimated)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks gestational age
  Number of ongoing pregnancies (defined as pregnancies passed beyond 12 weeks gestational age) divided by the number of women randomized

SECONDARY OUTCOMES:
Clinical pregnancy rate | 6 weeks after embryo transfer
  Number of clinical pregnancies (defined as presence of at least one intrauterine gestational sac with fetal pole and cardiac activity on TVS scan at 4-6 weeks after the ET) divided by the number of women randomized
Implantation rate | 6 weeks after embryo transfer
  Number of gestational sacs on TVS scan at 4-6 weeks after ET divided by the number of transferred embryos
Miscarriage rate | 12 weeks gestational age
  Number of first trimester miscarriages (before 12 weeks gestational age) divided by the number of clinical pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Gibreel, MD, Principal Investigator — Mansoura University; Mohamed S Abdelhafez, MD, Study Director — Mansoura University; Hasan El Maghraby, MD, Study Director — Alexandria University; Hamed Yossef, MD, Study Chair — Mansoura University
Locations (3):
- Egypt (3):
  - Fertility Care Unit (FCU) in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate
  - Department of Obstetrics and Gynecology, Alexandria
  - RAHEM Fertility Centre, Zagazig